CLINICAL TRIAL: NCT03269045
Title: An Open-label, Single-arm, Phase 2 Study of ORL-1B in Patients With Biotinidase Deficiency
Brief Title: Study of ORL-1B in Patients With Biotinidase Deficiency
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Orpha Labs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Biot-1
Record Dates: First submitted 2017-08-28; First posted 2017-08-31 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Biotinidase Deficiency
MeSH Terms: conditions — Biotinidase Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with ORL-1B. (Other): Pediatric patients with biotinidase deficiency.
  Interventions: Drug: ORL-1B

INTERVENTIONS:
Drug: ORL-1B — Oral ORL-1B

SUMMARY:
An Open-label, Single-arm, Phase 2 Study of Biotin in Patients With Biotinidase Deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of biotinidase deficiency.
* Less than 18 years old.

Exclusion Criteria:

* Diagnosis of any other disease that is not a manifestation of biotinidase deficiency.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2013-08-31 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Improvement in seizure frequency | 12 months
  Statistically significant improvement in seizure frequency after the ORL-1B treatment.

IPD SHARING:
Plan to Share IPD: No